CLINICAL TRIAL: NCT06057818
Title: Airway Ultrasound Versus Mallampati Score as a Predictor of Difficult Direct Laryngoscopy in Obese Patients an Observational Study
Brief Title: Airway Ultrasound Versus Mallampati Score as a Predictor of Difficult Direct Laryngoscopy in Obese Patients
Status: Recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sherif Hany Adly Loka, assistant lecturer, Ain Shams University
Other Study IDs: MD99/2023
Record Dates: First submitted 2023-09-20; First posted 2023-09-28 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Airway Ultrasound; Difficult Intubation; Mallampati Score

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to evaluate the ability of pre-operative ultrasound assessment of neck anatomy in predicting difficult laryngoscopy in obese patients undergoing elective surgery requiring tracheal intubation and comparing it to conventional methods as the Mallampati score in anticipating difficult laryngoscopy.

DETAILED DESCRIPTION:
All patients enrolled in the study will be consented by written and informed consent to do the airway ultrasound before induction.

During pre-anesthetic evaluation of the patients, demographic variables will be collected from each patient and clinical screening tests to predict difficult airway will be performed in the form of Mallampati score sitting in neutral position.

The patient will be admitted to the pre-anesthesia care unit, attended by anesthesiologist experienced in ultrasound.

The ultrasound will be done with the patients seated, head held in neutral position, using the linear probe 13-6i of SonoSite model M-Turbo c with 13-6Mega Hertz frequency, Preoperative ultrasonographic airway assessment will be performed for all patients in the study, Patients will be explained about the procedure before starting the study.

Operator will position himself on the right side of the patient, holding the ultrasound transducer in the right hand, the transducer will be placed transversely just above the suprasternal notch to visualize the tracheal cartilage, a horseshoe shaped hypoechoic structure, if tracheal deviation is present, the transducer might need to be moved laterally to locate the trachea and its position should be marked out with a pen, the transducer will be moved cephalad to inspect the remaining structures.

The probe will be placed in the transverse axis, ultrasound distances will be measured as the distance from the hyoid bone to skin surface, the distance from skin to anterior commissure of the vocal cords and the distance from skin to the trachea at the level of the suprasternal notch.

All measurements will be done using the ultrasound measure and pointing in mm, gain and depth will be adjusted accordingly to obtain best view.

Difficult intubation tray and settings will be available and ready before induction.

Patients will be taken to the operating room and will be monitored by American Society of Anesthesiologists standard monitors: ECG, noninvasive blood pressure, pulse oximetry, capnography then after pre-oxygenation with fraction of inspired oxygen : 100% for 3 min, intravenous (IV) midazolam 1 mg and fentanyl 1 µg/kg, anesthesia will be induced with injection of propofol 2 mg/kg. After muscle relaxation with injection of rocuronium 0.8 mg/kg IV and ventilation with oxygen and sevoflurane 1.5% for 3 min, direct laryngoscopy will be done by attending anesthesiologist (with more than 2 years of experience post-qualification) using an appropriate size curved Macintosh blade, and the modified Cormack-Lehane (CL) laryngoscopic grade will be evaluated and documented. The correct positioning of the endotracheal tube will be confirmed via capnography and bilateral auscultation of lungs.

The view of the glottis aperture will be assessed using the modified Cormack Lehane scale at which grading of 2b, 3 and 4 will be considered a difficult intubation view for the patient.

The intubating anesthesiologist will not be involved in preoperative clinical and sonographic airway assessment. Therefore, he will be blinded to the findings of preoperative airway evaluation.

Anesthesia will be maintained by sevoflurane, booster doses of rocuronium and fentanyl as needed.

Patients are assessed regarding:

* Mallampati score
* Distance from skin to vocal cords
* Distance from skin to anterior aspect of trachea at level of suprasternal notch
* Distance from skin to hyoid bone

ELIGIBILITY:
Inclusion Criteria:

1. Both sexes
2. Age from18 to 60 years old
3. With an American Society of Anesthesiologists physical status classification score of I to III,
4. Scheduled for elective surgical procedure requiring endotracheal intubation
5. Body mass index more than 30 kg/m2.

Exclusion Criteria:

1. Patient refusal
2. Emergency surgery
3. Patients with history of airway or neck surgery
4. Neck mobility abnormalities
5. Syndromatic patients
6. Pre-existing airway malformations or pathology like facial or cervical fractures, maxillofacial abnormalities, cervical tumors or goiter.
7. History of difficult intubation.
8. Patients with tracheostomy tubes.
9. Pregnant patients.
10. Body mass index less than 30 kg/m2.
11. ASA IV or above patients.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: patients of both sexes (18-60 years old) with an American Society of Anesthesiologists physical status classification score of I to III, scheduled for elective surgical procedure requiring endotracheal intubation and body mass index more than 30 kg/m2.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Comparison between the Mallampati score and the airway ultrasound | 6 months
  Comparison between the Mallampati score and the airway ultrasound measurements in the prediction of difficult intubation in obese patients

SECONDARY OUTCOMES:
comparison between each airway ultrasound measurement | 6 months
  The sensitivity and specificity of each airway ultrasound measurement to anticipate difficult intubation.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt